CLINICAL TRIAL: NCT07006506
Title: Phase II Open Label Prospective Nonrandomized Trial of Belumosudil for Switch-Maintenance Prophylaxis of Graft-versus-Host Disease in Allogeneic Hematopoietic Cell Transplantation
Brief Title: A Study of Belumosudil in People at Risk of Developing Graft-Versus-Host Disease After a Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-033
Record Dates: First submitted 2025-05-22; First posted 2025-06-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Graft Versus Host Disease; Graft Vs Host Disease; Hematologic Malignancy
Keywords: Graft Versus Host Disease; Graft Vs Host Disease; Hematologic Malignancy; Hematologic malignancy in morphologic remission; Belumosudil; Stem Cell Transplant; Memorial Sloan Kettering Cancer Center; 25-033
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with hematologic malignancy in morphologic remission (Experimental): Participants will be diagnosed with a hematologic malignancy in morphologic remission
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Belumosudil is an oral selective inhibitor of Rho-GTPase-associated coiled-coil kinase 2 (ROCK2)

SUMMARY:
The purpose of this study is to find out whether adding belumosudil to a usual approach for reducing the risk of graft-versus-host disease (GVHD) may be an effective GVHD prevention approach for people with blood cancer who have a stem cell transplant. The investigators will also look at the safety of the study approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years-old at time of consent.
* Diagnosis: hematologic malignancy in morphologic remission who will be treated with RI or NMA conditioning and GVHD prophylaxis CNI-based (CNI without PTCY) plus abatacept or PTCY-based (CNI with PTCY).
* Recipients of 7-8/8 related or unrelated HLA-matched or related haploidentical donor.
* Peripheral blood stem cell graft
* Allo-HCT day <120 at time of consent

Post-HCT inclusion criteria (within 3 weeks before start of belumosudil treatment)

* Patient has received an allo-HCT transplant and is in morphologic remission (blasts <5%, no evidence of extramedullary disease in AML or MDS). Patients with CR with incomplete count recovery (CRp or CRi) or minimal residual disease are allowed.
* Patient has achieved engraftment. Engraftment is defined as ANC≥500/μL and platelets ≥ 20000/μL on 3 consecutive measurements (each occurring at least 1 day apart). The patient must not have had a platelet transfusion within 7 days before the first measurement.
* Patient is ≥ 80 days and ≤ 20 days from allo-HCT infusion.
* Karnofsky score ≥ 70%.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3x upper limit of normal (ULN)
* Total bilirubin ≤1.5 x ULN (unless benign congenital hyperbilirubinemia).
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2
* Female subjects of childbearing potential (≤ 50 years old) have a negative serum or urine pregnancy test. Females of childbearing potential are defined as females without prior hysterectomy or who have had any evidence of menses in the past 12 months.

  ° Sexually active females of childbearing potential enrolled in the study must agree to consistently use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes: * Intrauterine device (IUD) plus one barrier method * Stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal) plus one barrier method * 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gel that contain a chemical to kill sperm); or * A vasectomized partner
* For male subjects who are sexually active and who are partners of females of childbearing potential: Agreement to use two forms of contraception as per above and to not donate sperm during the treatment period and for at least 3 months after the last dose of study drug.

Exclusion Criteria:

* Recipient of CD34+ selected or engineered stem cell graft.
* Treatment with in vivo T cell depletion (e.g. anti-thymocyte globulin).
* Evidence of current uncontrolled cardiovascular conditions, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Pulmonary dysfunction with DLCO <50% corrected for hemoglobin

Post-HCT exclusion criteria

* Uncontrolled infection, including active hepatitis B and C. Definitive therapy for infection is required and must have no signs of progression within 7 days of the first day of study drug treatment.
* Use of investigational agent within 14 days pre-HCT or anytime thereafter.
* Active acute or chronic GVHD requiring systemic therapy (topical or local therapies are allowed).
* Active treatment with corticosteroids at a dose of ≥ 0.25 mg/kg/day for non-GVHD indication.
* Uncontrolled psychosis, active suicidal ideation, or psychiatric hospitalization within the past year
* Female patient who is pregnant or breastfeeding.
* Prior therapy with belumosudil.
* Known allergy or sensitivity to belumosudil or any other ROCK2 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2029-05-21 (Estimated); Study Completion 2029-05-21 (Estimated)

PRIMARY OUTCOMES:
Change in GVHD/relapse-free survival (GRFS) at 1-year post-Hematopoietic Cell Transplantation (HCT) | 1 year
  The primary objective is to assess the efficacy of belumosudil in the improvement of GRFS at 1-year post-HCT for patients receiving PTCY GVHD prophylaxis and separately for participants receiving CNI-based (CNI without PTCY) plus abatacept GVHD prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ponce, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org